CLINICAL TRIAL: NCT03311529
Title: Effectiveness and Underlying Mechanisms of Applied Relaxation as Indicated Preventive Intervention in Subjects at Increased Risk for Mental Disorders
Brief Title: Effectiveness and Underlying Mechanisms of Applied Relaxation as Indicated Preventive Intervention
Acronym: EASY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Eva Asselmann, Study Principal Investigator, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AS 497/1-1
Record Dates: First submitted 2017-03-10; First posted 2017-10-17 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Anxiety Disorders; Depressive Disorder; Stress Disorder
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Applied Relaxation (Experimental)
  Interventions: Behavioral: Applied Relaxation
- usual care (No Intervention)

INTERVENTIONS:
Behavioral: Applied Relaxation — 10 training sessions (90 min. each) in Applied Relaxation (group format)
  Arms: Applied Relaxation

SUMMARY:
As mental disorders constitute a core health care challenge of the 21th century, increased research efforts on preventive interventions are indispensable. In the field of clinical psychology, indicated preventive interventions targeted to those with initial symptomatology appear particularly promising. Applied relaxation (AR) is a well-established intervention technique proven to effectively reduce tension/distress, anxiety and depressive symptoms in the context of treatment of a wide variety of manifest mental disorders as well as somatic illnesses. However, it has not been studied so far whether AR as indicated preventive intervention in subjects with initial symptomatology but no full-threshold mental disorder yet is capable to prevent a further symptom escalation. This randomized controlled trial in subjects with elevated tension/distress, anxiety or depressive symptomatology aims to investigate whether an AR intervention (10 sessions à 60 min) can (a) effectively reduce present psychopathological symptoms as well as (b) prevent a further symptom progression to full-threshold DSM-5 mental disorders. Putative mediators (physiological, emotional, cognitive and behavioral changes including heart rate and heart rate variability, hair and salivary cortisol secretion, affectivity, self-efficacy, internal locus of control and cognitive / behavioral coping) and moderators (sex, age, symptom severity at baseline and homework adherence during the intervention course) of the intervention/preventive efficacy will be additionally studied. Predictor and outcome measures will be assessed both conventionally (via personal interview, questionnaires and physiological measures during the respective main assessment) and with ecological momentary assessments (EMA, applied via smart phone over a 1-week interval following the respective main assessment) in everyday life.

ELIGIBILITY:
Inclusion criteria are as follows: at least mild symptoms of tension/distress, anxiety or depression (DASS-21 score of 8 or higher on tension/stress, of 4 or higher on anxiety, and of 5 or higher on depression)

Exclusion criteria are as follows: (1) a 12-month diagnosis of any mental disorder, (2) lifetime psychotic symptoms, (3) current psychological or psychopharmacological intervention, (4) acute suicidality

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 277 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
primary outcome intervention efficacy | from baseline- (immediately prior to the 10-week intervention) to post-assessment (immediately after completion of the 10-week intervention or a comparable time frame in controls)
  reduction of tension/distress, anxiety and depressive symptoms (DASS-21 tension/stress, anxiety and depression)
primary outcome prevention efficacy | from entry exam (prior to the 10-week intervention) to follow-up-assessment (12 months after completion of the 10-week intervention or a comparable time frame in controls)
  rates of incident mental disorders (first incidence or recurrence of sub-threshold or threshold DSM-5-defined mental disorders; DIA-X/CIDI)

SECONDARY OUTCOMES:
secondary outcomes intervention efficacy | from baseline- (immediately prior to the 10-week intervention) to post-assessment (immediately after completion of the 10-week intervention or a comparable time frame in controls)
  other symptom changes (DSM-5 CCSM anxiety, depression, anger, somatic symptoms, sleep disturbance)
secondary outcomes intervention efficacy | from baseline- (immediately prior to the 10-week intervention) to post-assessment (immediately after completion of the 10-week intervention or a comparable time frame in controls)
  other clinical changes from baseline- to post-assessment (e.g. impairment, disability)
secondary outcomes prevention efficacy | from post-assessment (immediately after completion of the 10-week intervention or a comparable time frame in controls) to follow-up-assessment (12 months after completion of the 10-week intervention or a comparable time frame in controls)
  changes of tension/distress, anxiety and depressive symptoms (DASS-21 tension/stress, anxiety and depression)
secondary outcomes prevention efficacy | from post-assessment (immediately after completion of the 10-week intervention or a comparable time frame in controls) to follow-up-assessment (12 months after completion of the 10-week intervention or a comparable time frame in controls)
  other symptom changes (DSM-5 CCSM anxiety, depression, anger, somatic symptoms, sleep disturbance)
secondary outcomes prevention efficacy | from post-assessment (immediately after completion of the 10-week intervention or a comparable time frame in controls) to follow-up-assessment (12 months after completion of the 10-week intervention or a comparable time frame in controls)
  other clinical changes (e.g. number of symptoms/diagnoses, impairment, disability)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Asselmann, PhD, Principal Investigator — Technische Universität Dresden
Locations (1):
- Technische Universität Dresden, Dresden, Germany

REFERENCES:
- [Derived] Asselmann E, Ruckert F, Kische H, Zenker M, Pieper L, Beesdo-Baum K. Cognitive, behavioral, and affective mechanisms underlying the efficacy of Applied Relaxation in reducing psychopathological symptoms: A randomized controlled trial. J Mood Anxiety Disord. 2024 Feb 22;6:100055. doi: 10.1016/j.xjmad.2024.100055. eCollection 2024 Jun. PMID 40655922
- [Derived] Asselmann E, Zenker M, Ruckert F, Kische H, Pieper L, Beesdo-Baum K. Ecological momentary assessment and applied relaxation: Results of a randomized indicated preventive trial in individuals at increased risk for mental disorders. PLoS One. 2023 Jun 8;18(6):e0286750. doi: 10.1371/journal.pone.0286750. eCollection 2023. PMID 37289760
- [Derived] Beesdo-Baum K, Zenker M, Ruckert F, Kische H, Pieper L, Asselmann E. Efficacy of Applied Relaxation as indicated preventive intervention in individuals at increased risk for mental disorders: A randomized controlled trial. Behav Res Ther. 2022 Oct;157:104162. doi: 10.1016/j.brat.2022.104162. Epub 2022 Jul 20. PMID 35930850
- [Derived] Kische H, Zenker M, Pieper L, Beesdo-Baum K, Asselmann E. Applied relaxation and cortisol secretion: findings from a randomized controlled indicated prevention trial in adults with stress, anxiety, or depressive symptoms. Stress. 2022 Jan;25(1):122-133. doi: 10.1080/10253890.2022.2045939. PMID 35285766